CLINICAL TRIAL: NCT00274885
Title: Study of the Relationship Between the Rate of Residual Platinum in the Blood and the Incidence of Persistent Neurotoxicity in Patients Treated for Gastrointestinal Cancer With Oxaliplatin
Brief Title: Relationship Between Platinum Levels in the Blood and Neurotoxicity in Patients Who Are Receiving Oxaliplatin for Gastrointestinal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454401; GERCOR-TAUROX; SANOFI-GERCOR-TAUROX; EU-20573
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2007-05

CONDITIONS: Cancer
Keywords: neurotoxicity; carcinoma of the appendix; recurrent anal cancer; stage I anal cancer; stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; stage IV anal cancer; localized extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; localized gallbladder cancer; recurrent gallbladder cancer; unresectable gallbladder cancer; recurrent gastric cancer; stage IV gastric cancer; recurrent colon cancer; recurrent rectal cancer; recurrent esophageal cancer; localized gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; gastrointestinal stromal tumor; advanced adult primary liver cancer; localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent small intestine cancer; small intestine adenocarcinoma; small intestine leiomyosarcoma; small intestine lymphoma; stage IV pancreatic cancer; metastatic extrahepatic bile duct cancer; metastatic gallbladder cancer; stage IA gastric cancer; stage IB gastric cancer; stage IIA gastric cancer; stage IIB gastric cancer; stage IIIA gastric cancer; stage IIIB gastric cancer; stage IIIC gastric cancer; stage I colon cancer; stage IIA colon cancer; stage IIB colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer; stage IVA colon cancer; stage IVB colon cancer; stage I rectal cancer; stage IIA rectal cancer; stage IIB rectal cancer; stage IIC rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer; stage IIIC rectal cancer; stage IVA rectal cancer; stage IVB rectal cancer; stage IA esophageal cancer; stage IB esophageal cancer; stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Neoplasms; Neurotoxicity Syndromes; Appendiceal Neoplasms; Anus Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Gastrointestinal Stromal Tumors; Carcinoma, Hepatocellular; Pancreatic Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Learning about the relationship between platinum levels in the blood and neurotoxicity in patients receiving oxaliplatin may help plan treatment and may help patients live more comfortably.

PURPOSE: This phase IV trial is studying the relationship between platinum levels in the blood and neurotoxicity in patients who are receiving oxaliplatin for gastrointestinal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the relationship between residual platinum levels in the blood and persistent neurotoxicity in patients receiving oxaliplatin for gastrointestinal cancer.

Secondary

* Determine the pharmacokinetics of oxaliplatin in these patients.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive oxaliplatin IV over 2 hours. Treatment repeats every 2-3 weeks in the absence of disease progression or unacceptable toxicity.

Neurological function and platinum levels in the blood are assessed at baseline, after each course of oxaliplatin, and at the end of study treatment.

PROJECTED ACCRUAL: A total of 58 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of gastrointestinal cancer
* Receiving or planning to receive 8 months of oxaliplatin-based chemotherapy
* No pre-existing neuropathy
* No CNS disease or cerebral metastases

PATIENT CHARACTERISTICS:

* WHO 0-1
* Life expectancy ≥ 12 weeks
* No biliary or gastro-duodenal obstruction
* No familial, social, geographical, or psychological condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other concurrent drug or agent that is potentially neurotoxic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2005-10

PRIMARY OUTCOMES:
Relationship between residual platinum levels in the blood and persistent neurotoxicity

SECONDARY OUTCOMES:
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lechat, Study Chair — CHU Pitie-Salpetriere
Locations (6):
- France (6):
  - CHU de Grenoble - Hopital Michallon, Grenoble
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Clinique Saint Jean, Lyon
  - Hopital Saint Antoine, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris